CLINICAL TRIAL: NCT01716949
Title: Multi-institutional Phase I/II Study: Neoadjuvant Chemoradiation With 5-FU (or Capecitabine) and Oxaliplatin Combined With Deep Regional Hyperthermia in Locally Advanced or Recurrent Rectal Cancer
Brief Title: Neoadjuvant Chemoradiation With 5-FU(or Capecitabine) and Oxaliplatin Combined With Hyperthermia in Rectal Cancer
Acronym: HyRec
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESHO201107/001
Record Dates: First submitted 2012-10-05; First posted 2012-10-30 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; recurrent rectal cancer; hyperthermia; radiation; chemoradiation; 5-FU; capecitabine; oxaliplatin
MeSH Terms: conditions — Rectal Neoplasms; Hyperthermia | interventions — Radiotherapy; Diathermy; Fluorouracil; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HyRec (Experimental): Radiotherapy, Hyperthermia, 5-Fluorouracil (may be replaced by Capecitabine), Capecitabine (may be replaced by 5-Fluorouracil), Oxaliplatin
  Interventions: Radiation: Radiotherapy; Procedure: Hyperthermia; Drug: 5-Fluorouracil; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Radiotherapy — 45 up to 50.4 Gy; daily dose 1,8 Gy, 5 days per weeks
Procedure: Hyperthermia — 10 sessions, therapeutic time 60 min
Drug: 5-Fluorouracil — 250 mg/m^2/d as continuous i.v. infusion on d1-14, 22-35 (may be preplaced by Capecitabine)
  Other Names: all brands of 5-Fluorouracil are allowed
Drug: Capecitabine — 1650 mg/m^2/d oral intake d1-14, 22-35 (may be replaced by 5-Fluorouracil)
  Other Names: all brands of Capecitabine are allowed
Drug: Oxaliplatin — 50 mg/m^2/d as 2-hour bolus infusion on d2, 9, 23, 30
  Other Names: all brands of oxaliplatin are allowed

SUMMARY:
This trial examines the feasibility, effectiveness and safety of a combination of radiotherapy (over a period of five weeks) and chemotherapy (with 5-FU or Capecitabine and Oxaliplatin) and 10 fractions of deep regional hyperthermia in patients with primary locally advanced or locally recurrent rectal cancer. Previous pelvic irradiation in case of a local recurrence is not excluded from the trial. The treatment protocol aims on a preoperatively improved tumor regression allowing less aggressive surgery in primary locally advanced rectal cancer and a higher rate of curative resections in heavily pretreated locally recurrent rectal cancers.

Primary endpoint of the trial is the feasibility rate of a multimodal regimen consisting of radiochemotherapy and hyperthermia. Secondary endpoints are local control, survival rates, and toxicity. It is planned to include a total number of 59 patients over a period of 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed, locally advanced or recurrent (any recurrence of tumor within the lesser pelvis; resectable or non-resectable) adenocarcinoma of the rectum (UICC stage IIB-IV); distant oligo-metastases may be present.
* ECOG-performance status < 2
* Sufficient bone marrow function:
* WBC > 3,5 x 10^9/l
* Neutrophil granulocytes > 1,5 x 10^9/l
* Platelets > 100 x 10^9/l
* Hemoglobin > 10 g/dl
* Sufficient liver function: Bilirubin < 2,0 mg%, SGOT, SGPT, alkaline phosphatase, gGT less than 3 times upper limit of normal
* Serum creatinine < 1,5 mg%, glomerular filtration rate (or comparable test) > 50 ml/min
* Signed study-specific consent form prior to therapy
* Fertile patients must use effective contraception during and for 6 months after study treatment
* Considered fit for oxaliplatin and 5-FU-containing combination chemotherapy

Exclusion Criteria:

* Pelvic radiotherapy during the last 12 months
* Pregnant or lactating/nursing women
* Drug addiction
* On-treatment participation on other trials
* Active intractable or uncontrollable infection
* Prior or concurrent malignancy (≤ 5 years prior to enrolment in study) except rectal cancer or non-melanoma skin cancer or cervical carcinoma FIGO stage 0-1 if the patient is continuously disease-free
* Chronic diarrhea (> NCI CTC-Grad 1)
* Chronic inflammatory disease of the intestine
* Collagen vascular disease
* The presence of congenital diseases with increased radiation sensitivity, for example teleangiectatic ataxia, or similar
* Pre-existing uncontrolled cardiac disease, signs of cardiac failure, or rhythm disturbances requiring therapy
* Myocardial infarction within the past 12 months
* Congestive heart failure
* Complete bundle branch block
* New York Heart Association (NYHA) class III or IV heart disease
* Known allergic reactions on study medication
* Cardiac pacemaker
* Disease that would preclude chemoradiation or deep regional hyperthermia
* Any metal implants (with exception of non-clustered marker clips)
* Psychological, familial, sociological, or geographical condition that would preclude study compliance
* Patients deemed technically unsatisfactory for deep regional hyperthermia
* Cardiac symptoms (> NCI CTCAE Grade 1) due to pretreatment with fluoropyrimidines
* Neurological symptoms (> NCI CTCAE Grade 1) due to pretreatment with oxaliplatin
* Rare hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2012-09; Primary Completion 2022-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Feasibility rate (i.e. rate of patients not experiencing dose-limiting toxicity [DLT]) | Participants will be followed for the duration of therapy and for 6 weeks after the last study treatment dose (approximately 11 to 12 weeks)
Number of hyperthermia applications by patient | Duration of therapy (approximately 5 to 6 weeks)

SECONDARY OUTCOMES:
Local progression-free survival | Participants will be followed for up to 5 years after the end of therapy (Follow up period)
Distant metastasis-free survival | Participants will be followed for up to 5 years after the end of therapy (Follow up period)
Overall survival | Participants will be followed for up to 5 years after the end of therapy (Follow up period)
Response rate | Participants will be followed for up to 5 years after the end of therapy (Follow up period)
Rate of R0-resections | Only of participants who are considered as resectable receive surgery in curative intention 4-6 weeks after completion of chemoradiation (results app. after 10 to 12 weeks after start of therapy)
Rate of acute and late toxicity | Participants will be followed for up to 5 years after the end of therapy (Follow up period)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Ott, MD, Principal Investigator — Strahlenklinik, Universitätsklinikum Erlangen
Locations (6):
- Germany (6):
  - Klinik Bad Trissl, Innere Medizin, Bad Trissl
  - University Hospital, Düsseldorf
  - Universitätsklinikum Erlangen, Strahlenklinik, Erlangen
  - LMU München, Campus Großhadern, Medizinische Klinik III, Hyperthermie, München
  - Schlossbergklinik, Oberstaufen
  - Universitätsklinikum Tübingen, Radioonkologie, Tübingen

REFERENCES:
- [Derived] Ott OJ, Gani C, Lindner LH, Schmidt M, Lamprecht U, Abdel-Rahman S, Hinke A, Weissmann T, Hartmann A, Issels RD, Zips D, Belka C, Grutzmann R, Fietkau R. Neoadjuvant Chemoradiation Combined with Regional Hyperthermia in Locally Advanced or Recurrent Rectal Cancer. Cancers (Basel). 2021 Mar 13;13(6):1279. doi: 10.3390/cancers13061279. PMID 33805731